CLINICAL TRIAL: NCT06902701
Title: Endoscopic Submucosal Dissection vs. Transanal Endoscopic Surgery for Rectal Neoplasia: A Multicenter Prospective Observational Cohort Study
Brief Title: Endoscopic Submucosal Dissection vs. Transanal Endoscopic Surgery for Rectal Neoplasia
Acronym: ESTER
Status: Not yet recruiting | Type: Observational
Sponsor: Turkish Society of Colon and Rectal Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: TKRCD2
Record Dates: First submitted 2025-03-16; First posted 2025-03-30 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Rectal Neoplasms
Keywords: endoscopic submucosal dissection; transanal endoscopic surgery; early rectal neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Endoscopic Mucosal Resection; Transanal Endoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic submucosal dissection (ESD): Patients who underwent excision with endoscopic submucosal dissection
  Interventions: Procedure: Endoscopic Submucosal Dissection (ESD)
- Transanal endoscopic surgery (TES): Patients who underwent excision with transanal endoscopic surgery
  Interventions: Procedure: Transanal Endoscopic Surgery (TES)

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection (ESD) — Endoscopic excision of the rectal lesion by submucosal injection and circumferential mucosal incision using an electrosurgical knife with en-bloc resection intent
  Groups: Endoscopic submucosal dissection (ESD)
Procedure: Transanal Endoscopic Surgery (TES) — Transanal endoscopic surgery procedures include Transanal Minimally Invasive Surgery (TAMIS) and Transanal Endoscopic Operation (TEO). TAMIS will be performed using a single-port transanal access platform with standard laparoscopic instruments, including a high-definition camera, an insufflation system, and endoscopic graspers. The lesion will be circumferentially excised using electrocautery or an energy device, ensuring full-thickness resection when necessary. The defect will be managed based on its size, with primary closure using absorbable sutures or left to heal by secondary intention. TEO will be conducted using a rigid transanal endoscopic platform with a stereoscopic optical system to enhance visualization. The lesion will be marked, and a full-thickness or submucosal excision will be performed using endoscopic instruments and electrosurgical devices. Post-resection, the rectal wall defect will be assessed, and primary closure will be performed when indicated to minimize post
  Groups: Transanal endoscopic surgery (TES)

SUMMARY:
This prospective observational cohort study aims to compare the clinical and procedural outcomes of Endoscopic Submucosal Dissection (ESD) and Transanal Minimally Invasive Surgery (TAMIS) for the treatment of early-stage rectal neoplasia. The study will evaluate recurrence rates, en bloc resection rates, R0 resection rates, procedure time, complication rates, and length of hospital stay over a 1-year follow-up period. Data will be collected from patients treated at multiple centers with expertise in ESD and TAMIS.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignancies globally, with early-stage rectal neoplasms being increasingly diagnosed due to widespread screening programs. This trend has led to a greater focus on organ-preserving treatment options, with endoscopic submucosal dissection (ESD) and transanal endoscopic surgery (TES) emerging as key techniques for local excision. ESD allows for en bloc resection of superficial lesions with high histological completeness but has a steep learning curve and a higher perforation risk. In contrast, TES, performed using transanal minimally invasive surgery (TAMIS) or transanal endoscopic operation (TEO), facilitates full-thickness excision and is more commonly used in Western surgical practice.

Each technique presents unique advantages and challenges. ESD is minimally invasive, preserves rectal function, and reduces postoperative complications such as fecal incontinence. However, its prolonged procedure time and technical difficulty limit its widespread adoption. TES, utilizing standard laparoscopic instruments, offers superior visualization and facilitates excision of deeper lesions but may lead to rectal wall defects, increased postoperative pain, and anorectal dysfunction. While studies suggest similar en bloc and recurrence rates between the two methods, discrepancies exist in procedural efficiency, hospital stay, and morbidity rates, with ESD potentially offering a shorter hospitalization period in certain cases.

Despite the increasing use of ESD and TES, a clear consensus on the optimal approach for early rectal neoplasms remains lacking. Existing data, primarily from high-volume centers in Asia, may not be fully applicable to Western populations. To address these gaps, this study aims to conduct a prospective, multi-center observational comparison of ESD and TES, assessing key outcomes such as recurrence rates, resection quality, complications, and hospital stay. The findings will contribute to refining treatment strategies and improving clinical decision-making for rectal neoplasm management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Non-pedunculated (sessile) lesions larger than 2 cm.
* Lesions located within 15 cm from the anal verge confirmed by sigmoidoscopy or magnetic resonance imaging (MRI)

Exclusion Criteria:

* Evidence of lymph node involvement, T2 rectal tumors, or distant metastasis on preoperative imaging modalities (MRI, ERUS, CT)
* Previous attempt at endoscopic resection
* Previous rectal surgery
* Previous pelvic radiation therapy
* Inflammatory bowel diseases (Crohn's disease, Ulcerative colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rectal neoplasia undergoing treatment with either ESD or TES at participating centers. Patients will be assigned to ESD or TES based on physician preference, patient choice, and institutional availability.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | Immediately post-procedure.
  Proportion of patients with histologically confirmed tumor-free margins. All pathological evaluations will be performed according to the College of American Pathologists (CAP) protocol (version 4.3.0.0, 2023)
Recurrence Rate | 12 months post-procedure.
  Proportion of patients with tumor recurrence at follow-up endoscopy within 12 months, histologically confirmed from resected visible residual disease or, if absent, from scar biopsies.

SECONDARY OUTCOMES:
En Bloc Resection Rate | Immediately post-procedure.
  Proportion of patients where the tumor was removed in a single piece. All pathological evaluations will be performed according to the College of American Pathologists (CAP) protocol (version 4.3.0.0, 2023)
Procedure Time | Immediately post-procedure.
  Total duration of the procedure (minutes).
Complication Rate | Up to 30 days post-procedure.
  Incidence of adverse events, including all intraoperative and postoperative according to Clavien-Dindo classification.
Length of Hospital Stay | Perioperative/Periprocedural
  Duration of hospitalization (days).
Fecal Incontinence | Pre-procedure and within the first 12 months post-procedure.
  Patient-reported outcomes will be assessed using the Wexner Incontinence Score, a validated instrument that quantifies the frequency and severity of fecal incontinence. Scores range from 0 (perfect continence) to 20 (complete incontinence), with higher scores indicating greater dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Feza Karakayali, MD, Study Chair — Baskent University
Locations (5):
- Turkey (Türkiye) (5):
  - Private Office, Istanbul
  - Baskent University, Istanbul
  - Memorial Sisli Hospital, Istanbul
  - Dokuz Eylul University, Izmir
  - Acibadem Kent Hospital, Izmir

IPD SHARING:
Plan to Share IPD: Yes
There will be sharing of de-identified individual participant data (IPD) about both the primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available to qualified researchers upon reasonable request, starting 6 months after publication of the study results and for up to 5 years.
Access Criteria: Data will be shared via a secure data repository, and access will require an approved data-sharing agreement.
URL: https://arastirma.tkrcd.org.tr

REFERENCES:
- [Background] de Sousa IVG, Bestetti AM, Cadena-Aguirre DP, Kum AST, Mega PF, da Silva PHVA, Miyajima NT, Bernardo WM, de Moura EGH. Comparison of endoscopic submucosal dissection and transanal endoscopic surgery for the treatment of rectal neoplasia: A systematic review and meta-analysis. Clinics (Sao Paulo). 2025 Mar 13;80:100613. doi: 10.1016/j.clinsp.2025.100613. eCollection 2025. PMID 40086369
- See also: Related Info — https://arastirma.tkrcd.org.tr